CLINICAL TRIAL: NCT01818687
Title: A Multi-centre, Open-label Study Evaluating the Safety and Tolerability of Colestilan (MCI-196) in Paediatric Subjects With Chronic Kidney Disease Stages 3b to 5 and With Hyperphosphataemia Not on Dialysis
Brief Title: Safety and Tolerability Study of MCI-196
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study has been terminated because of insufficient patient recruitment.
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCI-196-E16
Record Dates: First submitted 2013-03-18; First posted 2013-03-26 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Kidney Disease; Not on Dialysis; Hyperphosphatemia; Paediatric
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — cholebine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MCI-196 (Flexible dose) (Experimental): MCI-196 BSA eq 3g, 6g, 9g, 12g or 15g
  Interventions: Drug: colestilan

INTERVENTIONS:
Drug: colestilan — body surface area equivalent (BSAeq) 3 g/day, 6 g/day, 9 g/day, 12 g/day or 15 g/day
  Other Names: BindRen

SUMMARY:
The objective of this study is to assess the safety and tolerability of colestilan (MCI-196) in paediatric subjects (aged 2 years to <18 years) with CKD stages 3b to 5, diagnosed with hyperphosphataemia, who are not on dialysis.

DETAILED DESCRIPTION:
This study has been terminated because of insufficient patient recruitment. There were no safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 years to <18 years with CKD stages 3b to 5, not on dialysis (stage 3b is defined as a glomerular filtration rate below 45 mL/min/1.73 m²).
* The subject has a documented diagnosis of hyperphosphataemia, as demonstrated by serum phosphorus (P) levels above the age-related upper limit of normal (ULN) (Kidney Disease Outcomes Quality Initiative [KDOQI] Clinical Practice Guidelines for Nutrition in Children with CKD updated 2008).
* The subject is on a stable P diet at baseline (as judged by the Investigator).

Inclusion criteria for subjects not currently treated with phosphate binders:

* The subject, with serum P not controlled despite being on an appropriate P diet, must demonstrate serum P levels >1.5 standard deviation (SD) above the KDOQI 2008 age-related mean value at any time during the screening period. Such subjects do not require wash-out and should proceed to baseline for the next visit if additional screening visits are not required.

Baseline inclusion criteria for subjects treated with phosphate binders:

* The subject must enter the wash-out period, during which he/she must demonstrate serum P levels >1.5 SD above the KDOQI 2008 age-related mean value at any time during the wash-out period (after stopping phosphate binders), and;
* The subject must demonstrate an increase in serum P levels by at least 10% above the pre wash-out level (after stopping phosphate binders).

Note: should a subject fail to meet any of the above criteria, the subject is permitted to be re-screened once after an interval of at least three months.

Exclusion Criteria:

* The subject has been diagnosed with hypocholesterolaemia (i.e., cholesterol levels below age-related normal ranges, per local practices)
* The subject has current clinically significant medical comorbidities, which may substantially compromise subject safety, or expose him/her to undue risk, or interfere significantly with study procedures and which, in the opinion of the Investigator, make the subject unsuitable for inclusion in the study (e.g., the subject currently has or has had a history of seizure disorders, dysphagia, swallowing disorders, predisposition to or current bowel obstruction, ileus or gastrointestinal [GI] disorders such as chronic or severe constipation [as judged by the Investigator], intestinal stenosis, intestinal diverticulum, sigmoid colitis, GI ulcers, current or a history of GI bleeding, or major GI tract surgery)
* The subject cannot stop treatment (prescription or over the-counter) of any of the following orally taken medications during the wash-out period: any product containing calcium (Ca), magnesium (Mg), aluminium compounds, sevelamer, lanthanum, ketosteril
* The subject is receiving immunosuppressant treatment for any medical condition at the baseline visit or is expected to receive such treatment during the course of the study
* The subject is considered as unstable on his/her current treatment for CKD within one month prior to screening (e.g., subjects starting treatment with vitamin D or its analogues, or other agents/procedures that may influence bone mineral metabolism [i.e, serum P and Ca levels]

Exclusion criteria for subjects treated with phosphate binders:

* The subject was treated with a combination of two or more phosphate binders within one month prior to screening

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who, due to hyperphosphataemia, require rescue treatment and/or discontinuation of therapy with colestilan. | 17 weeks

SECONDARY OUTCOMES:
Incidence of TEAEs of hypercalcaemia and hypocalcaemia | 17 weeks
Laboratory safety assessments | 17 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site, London, United Kingdom